CLINICAL TRIAL: NCT04356807
Title: Effect of Physiotherapy on the Promotion of Bone Mineralization in Preterm Infants
Brief Title: Physical Therapy to Prevent Osteopenia in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galaad Torró Ferrero (Other)
Responsible Party: Sponsor-Investigator, Galaad Torró Ferrero, Principal Investigator, Universidad de Murcia
Organization: Universidad de Murcia (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Fisio-Osteopenia
Record Dates: First submitted 2020-03-17; First posted 2020-04-22 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Metabolic Bone Disease
Keywords: Premature Infant; Physical Therapy Modalities
MeSH Terms: conditions — Bone Diseases, Metabolic; Premature Birth | interventions — Massage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Care Provider and Outcomes Assessor are masked to the objectives of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reflex Locomotion Therapy (Experimental): during 15 minutes once a day five days a week
  Interventions: Procedure: Reflex Locomotion Therapy
- Passive Joint Mobilizations (Experimental): during 15 minutes once a day five days a week
  Interventions: Procedure: Passive Joint Mobilizations
- Massage (Placebo Comparator): during 15 minutes once a day five days a week
  Interventions: Procedure: Massage

INTERVENTIONS:
Procedure: Reflex Locomotion Therapy — The exercises corresponding to the motor complexes of the 1st phase of the rolling reflex and the original creeping reflex were performed, dedicating one minute to each side and performing two repetitions in each session.
  Arms: Reflex Locomotion Therapy
Procedure: Passive Joint Mobilizations — Passive Joint Mobilizations with articular pressure described by Moyer-Mileur, et al. 1995 and modified by Vignochi, et al. 2008
  Arms: Passive Joint Mobilizations
Procedure: Massage — Soft massage with soft pressures in limbs, tactile stimulation and no motion.
  Arms: Massage

SUMMARY:
To determine whether reflex locomotion therapy is effective for the prevention of osteopenia in preterm infants and compare its effectiveness over other physiotherapeutic methods like passive joint mobilizations and massage

DETAILED DESCRIPTION:
Premature infants have smaller and low bone mineralization compared with term infants bones, since 80% of calcium uptake occurs at the end of pregnancy. Passive Physiotherapy has been effective in the treatment of osteopenia. Active mobilizations implemented by the baby itself, may be more effective than passive, as they cause muscle contraction from the Central Nervous System (CNS). Reflex locomotion therapy (RLT), stimulates CNS causing muscle contraction so it may be effective in the treatment of osteopenia in premature.

Objectives: To determine whether RLT is effective for the prevention of osteopenia in preterm infants and compare its effectiveness over other physiotherapeutic methods.

Methodology: Our study is a multicentre randomized clinical trial, with 90 children less than 34 weeks of gestational age, divided into three treatment groups, one will receive RLT, another will be treated with passive joint mobilizations with articular pressure; and last one will be done massage techniques. The treatment will last for one month, for the three groups. We intend to measure changes in mineralization, bone formation, and bone resorption, and anthropometry.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants
* 26 to 34 weeks of gestational age
* Admitted in neonates
* Hemodynamically stable
* Complete enteral nutrition
* Parents or guardians signed an informed consent authorizing the participation of the baby in this study.

Exclusion Criteria:

* Neurological disorders
* Mechanical ventilation

  * Bronchopulmonary dysplasia
* Congenital malformations
* Metabolic diseases
* Genetic diseases
* Intraventricular hemorrhage III-IV,
* Diuretic medication or corticosteroids
* Bone fractures at the time of inclusion.

Max Age: 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Change in Tibial Speed of Sound | Change measurement: Pre treatment (baseline), at two weeks of treatment and after four weeks of treatment (end of the treatment)
  In order to measure bone mineralization, we used the tibial sound velocity test, using for that purpose a quantitative ultrasound device. It was measured on the left tibia in its lower third, while keeping the knee flexed at a 90 degree angle. The measurement point was made perpendicular to the direction of the bone. Three to five consecutive measurements were made, after which the average of these measurements was calculated to have one unique measure in m/s.
Change in Serum biomarkers of Bone-specific phosphatase markers | Change measurement: Pre treatment (baseline), and after four weeks of treatment (end of the treatment)
  N-telopeptides from collagen bonds from serum
Change in Serum biomarkers of osteocalcin markers | Change measurement: Pre treatment (baseline), and after four weeks of treatment (end of the treatment)
  osteocalcin markers
Change in Serum biomarkers of Beta-cross Laps. | Change measurement: Pre treatment (baseline), and after four weeks of treatment (end of the treatment)
  Beta-cross Laps.
Change in Urine biomarkers of N-telopeptides from collagen bonds | Change measurement: Pre treatment (baseline), at two weeks of treatment and after four weeks of treatment (end of the treatment)
  N-telopeptides from collagen bonds

SECONDARY OUTCOMES:
Change in Height | Change measurement: Pre treatment (baseline), at two weeks of treatment and after four weeks of treatment (end of the treatment)
  For anthropometry, height in cm were collected
Change in Weight | Change measurement: Pre treatment (baseline), at two weeks of treatment and after four weeks of treatment (end of the treatment)
  measurements of weight in grams were collected
Change in Head circumference | Change measurement: Pre treatment (baseline), at two weeks of treatment and after four weeks of treatment (end of the treatment)
  For anthropometry, measurements of head circumference in cm were collected

CONTACTS AND LOCATIONS:
Overall Officials: Galaad Torró-Ferrero, MSc, Principal Investigator — Universidad de Murcia
Locations (3):
- Spain (3):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Torrecárdenas de Almería, Almería
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared after contacting the authors
Supporting Information: Study Protocol, ICF, CSR
Time Frame: indefinitive
Access Criteria: Data will be shared after contacting the authors under reasonable request

REFERENCES:
- [Background] Vignochi CM, Miura E, Canani LH. Effects of motor physical therapy on bone mineralization in premature infants: a randomized controlled study. J Perinatol. 2008 Sep;28(9):624-31. doi: 10.1038/jp.2008.60. Epub 2008 Jul 17. PMID 18633420
- [Background] Vignochi CM, Silveira RC, Miura E, Canani LH, Procianoy RS. Physical therapy reduces bone resorption and increases bone formation in preterm infants. Am J Perinatol. 2012 Sep;29(8):573-8. doi: 10.1055/s-0032-1310520. Epub 2012 Jul 6. PMID 22773291
- [Background] Moyer-Mileur L, Luetkemeier M, Boomer L, Chan GM. Effect of physical activity on bone mineralization in premature infants. J Pediatr. 1995 Oct;127(4):620-5. doi: 10.1016/s0022-3476(95)70127-3. PMID 7562289
- [Background] Shaw SC, Sankar MJ, Thukral A, Natarajan CK, Deorari AK, Paul VK, Agarwal R. Assisted Physical Exercise for Improving Bone Strength in Preterm Infants Less than 35 Weeks Gestation: A Randomized Controlled Trial. Indian Pediatr. 2018 Feb 15;55(2):115-120. Epub 2017 Dec 14. PMID 29242413
- [Background] Giannantonio C, Papacci P, Ciarniello R, Tesfagabir MG, Purcaro V, Cota F, Semeraro CM, Romagnoli C. Chest physiotherapy in preterm infants with lung diseases. Ital J Pediatr. 2010 Sep 26;36:65. doi: 10.1186/1824-7288-36-65. PMID 20868518
- [Background] El-shaarawy MK, Rahman SAA, Fakher M, El A, Salah WM. Effect of rolling on oxygen saturation and incubation period in preterm neonates with respiratory distress syndrome. Int J Dev Res. 2017;07(01):11319-11323.
- [Background] Sanz-Esteban I, Calvo-Lobo C, Rios-Lago M, Alvarez-Linera J, Munoz-Garcia D, Rodriguez-Sanz D. Mapping the human brain during a specific Vojta's tactile input: the ipsilateral putamen's role. Medicine (Baltimore). 2018 Mar;97(13):e0253. doi: 10.1097/MD.0000000000010253. PMID 29595683
- [Derived] Torro-Ferrero G, Fernandez-Rego FJ, Aguera-Arenas JJ, Gomez-Conesa A. Effect of physiotherapy on the promotion of bone mineralization in preterm infants: a randomized controlled trial. Sci Rep. 2022 Jul 8;12(1):11680. doi: 10.1038/s41598-022-15810-6. PMID 35804078
- [Derived] Torro-Ferrero G, Fernandez-Rego FJ, Jimenez-Liria MR, Aguera-Arenas JJ, Pinero-Penalver J, Sanchez-Joya MDM, Fernandez-Berenguer MJ, Rodriguez-Perez M, Gomez-Conesa A. Effect of physical therapy on bone remodelling in preterm infants: a multicenter randomized controlled clinical trial. BMC Pediatr. 2022 Jun 24;22(1):362. doi: 10.1186/s12887-022-03402-2. PMID 35739544

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT04356807/Prot_SAP_000.pdf